CLINICAL TRIAL: NCT01467180
Title: Myoglobin Reduction by High Cut-off (HCO) Continuous Veno- Venous Hemodialysis (CVVHD) in Patients With Rhabdomyolysis and an Increased Risk for Acute Kidney Injury
Brief Title: Myoglobin Removal by High Cut-off CVVHD
Acronym: HicoRhabdo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Dialysatoren GmbH (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1490; CIV-11-06-000843 (Other: Eudamed)
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Rhabdomyolysis; Renal Failure
Keywords: septeX; CVVH; CVHD; myoglobin
MeSH Terms: conditions — Rhabdomyolysis; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCO CVVHD (Experimental): treatment of rhabdomyolysis pts with septeX dialyzer
  Interventions: Device: septeX
- HF CVVH (Active Comparator): treatment of rhabdomyolysis pts with standard high flux dialyzer
  Interventions: Device: HF CVVH

INTERVENTIONS:
Device: septeX — continuous veno-venose hemodialysis (CVVHD) with dialysate flow rate (Qd)of 35ml/kg/h for 48h
  Arms: HCO CVVHD
Device: HF CVVH — continuous veno-venose hemofiltration (CVVH) with 35ml/kg/h UF-rate for 48h
  Arms: HF CVVH

SUMMARY:
A high cut-off dialyzer (septeX) is tested for the removal of myoglobin which is not efficiently removed by standard high flux dialysis membranes. Hypothesis: The high cut-off dialyzer (septeX) can remove 2-fold more efficiently myoglobin from the circulation of Rhabdomyolysis patients as by conventional treatment with standard high flux dialyzer.

DETAILED DESCRIPTION:
Excess myoglobin in the circulation is a causative pathogenetic factor of rhabdomyolysis associated with acute kidney injury (AKI). The rapid elimination of myoglobin by standard dialysis membranes is limited to its molecular weight of 17.8kDa, although some removal can be achieved when a convective therapy is applied.

Significant clearance for myoglobin has been reported for high flux membranes from < 8 mL/min (5) up to 22 mL/h (CVVH) (10) and for high cut-off (HCO) membranes a mean clearance rate of 36.2 mL/min in HD mode (7) and 39.2 mL/h in CVVH mode (5). The use of high cut-off (HCO) continuous veno- venous hemodialysis (CVVHD) may constitute a novel therapeutic strategy for effectively reduction of myoglobin in the patient's serum to ameliorate the course of AKI.

Previously, a case study of the removal of myoglobin by HCO-CVVH in one single patient with severe rhabdomyolysis was published.

ELIGIBILITY:
Inclusion Criteria:

* Acute Rhabdomyolysis
* placed central venous catheter
* Indication for RRT due to Serum CK level > 5000 u/L
* Age ≥ 18 years
* Signed ICF

Exclusion Criteria:

* End stage CKD (dialysis dependent) renal failure before manifestation of rhabdomyolysis
* Pregnancy or lactation
* Palliative treatment
* Participation in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Myoglobin plasma level | 24h
  Two fold- increased reduction of myoglobin plasma level in favor of the HCO CVVHD group compared with standard therapy group (HF-CVVH and fluid therapy, respectively) after 48 hours treatment time.

SECONDARY OUTCOMES:
eGFR | at 3 and 6 month after treatment
  Estimation of kidney function by estimated glomerular filtration rate (eGFR)
Duration of hospital stay (days)and Duration of ICU stay (days) | 6 month
Duration of dialysis dependence (days) | 6 month
Diuresis / oliguria (<0.5 ml/kg/12h)/ anuria | 6 month
patient survival | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Anästhesiologie, Intensivmedizin, Uni-Klinikum, Frankfurt am Main, Hesse, Germany